CLINICAL TRIAL: NCT06693739
Title: Regenerative Ability of Immature Necrotic Permanent Teeth Using Different Scaffolds (A Randomized Clinical Trial)
Brief Title: Regenerative Ability of Immature Necrotic Permanent Teeth Using Different Scaffolds
Acronym: regeneration
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mai Osama, Principal investigator, Teaching assistant, Endodontic department, Faculty of dentistry, Ainshams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 072030
Record Dates: First submitted 2024-11-13; First posted 2024-11-18 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Regeneration
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- no scaffold (Active Comparator): initiate bleeding using hand files size beyond apex with sharp strokes
  Interventions: Procedure: no scaffold
- platelets rich fibrin (Experimental): PRF is used as Scaffold by placing the compressed PRF membrane into canal
  Interventions: Procedure: Platelet rich fibrin
- hyaluronic acid (Experimental): hyaluronic acid will be delivered by syringe into canal
  Interventions: Procedure: hyaluronic acid

INTERVENTIONS:
Procedure: Platelet rich fibrin — PRF membrane is placed as a scaffold inside the canal with no hyaluronic acid
  Arms: platelets rich fibrin
Procedure: hyaluronic acid — hyaluronic acid gel is placed as a scaffold inside the canal with no PRF
  Arms: hyaluronic acid
Procedure: no scaffold — initiate bleeding using hand files size beyond apex with sharp strokes with no PRF or hyaluronic acid placed
  Arms: no scaffold

SUMMARY:
The goal of this clinical trial is to compare effect of different scaffolds on the regenerative potential of young permanent immature teeth with necrotic pulp. The main question it aims to answer is:

is there difference in regenerative potential using Hyaluronic acid and platelets rich fibrin as scaffolds in permanent immature teeth with necrotic pulp? participants will undergo regeneration protocol including hyaluronic acid and platelets rich fibrin as scaffolds Researchers will compare [hyaluronic acid , platelets rich fibrin , and no scaffold ] to see the regenerative potential

DETAILED DESCRIPTION:
The study will be conducted on 30 maxillary anterior teeth with open apex; with 10 maxillary anterior teeth with open apex in each group (n=10). The patient will be asked to pick an opaque sealed envelope that will contain a number from 1 to 3. The resultant number will determine in which group the participants will be placed. single blinding will be maintained in this study as the Outcomes Assessor and the patients will not be aware of their group/used scaffold Group (I) control group with no scaffold used. Group (II) using platelets rich fibrin ( PRF) as a scaffold. Group (III) using hyaluronic acid (HYA) as a scaffold.

Procedural steps:

1st visit

1.Patients will be given anesthesia with vasoconstrictor . rubber dam isolation and access will be done 2. gentle irrigation with 1.5-3% sodium hypochlorite (NaOCl) (20ml/5 mins) using needle with closed end and side-vents with needle placed 1mm from apex will be done 3.then, irrigation will be done with saline or 17% Ethylenediaminetetraacetic acid (EDTA) (20 mL/canal, 5 min) 4. The canal space will be dried using sterile paper points 5.1ml of calcium hydroxide (metapaste) will be delivered into canal space 6.Sterile cotton pellet will be inserted and access cavity will be sealed using 3-4mm of temporary restoration (Coltosol F; Coltene Whaledent, Altstatten, Switzerland) for 3 weeks.

2nd visit

1. Final visit for three groups will be scheduled when tooth is asymptomatic with no signs of discharge.
2. In case of persistent infection one or more visits will be scheduled for discharge and disinfection.
3. patient will be anesthetized using 3% mepivacaine without vasoconstrictor, proper isolation will be done, the temporary restoration and cotton pellet will be removed.
4. Canal will be irrigated using 17% EDTA (20ml/5mins).
5. Canals will be dried using sterile paper points.
6. In group (I) A sterile hand file size #50 will be used sharp strokes 2 mm beyond apex into the periapical tissue until bleeding is evident in cervical portion of canal In group (II) For the PRF preparation, 10Ml of the patient's whole blood will be collected in sterile tubes from the cubital vein. The tubes will be centrifuged for 10 minutes with a speed of 3000 rpm .

   Inside each test tube three layers will be formed: a base layer containing erythrocytes, an intermediate layer of PRF clot, and a surface layer of acellular plasma. The PRF clot will be separated from the other layers and then compressed in a PRF box (Intra-Lock International).

   The compressed PRF membrane will be rolled over itself to allow its implantation into the canal .

   The PRF membrane will be inserted inside the root canal and condensed apically with an endodontic hand plugger.

   In group (III)A sterile hand file size #50 will be used sharp strokes 2 mm beyond apex into the periapical tissue until bleeding is evident in cervical portion of canal then, hyaluronic acid hydrogel will be inserted inside the canal
7. MTA plug orifice plug as a capping material will be used to seal canal orifice.
8. 3-4 mm layer of glass ionomer (e.g. Fuji IX™, GC America, Alsip, IL) will be flowed gently over the capping material and light-cured for 40 s to seal the access cavity.
9. A postoperative standardized periapical radiograph will be taken for baseline records
10. After treatment is done patient will be recalled for follow-up every three months for one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age range from 9-20 years with no sex predilection. Systemically healthy patients.
* Non-vital maxillary anterior presenting with or without signs and/or symptoms of periapical pathology.
* No mobility.
* Pocket depth less than 3 mm.

Exclusion Criteria:

* Teeth with vertical fracture
* Periodontal involved teeth and non-restorable teeth
* Lack of patient cooperation

Ages: 9 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Clinically by absence of pain and/or swelling | 1 year
  absence of pain is measured clinically by absence of pain in response to percussion and palation in relation to the related tooth
absence or change of periapical radiolucency. | 1 year
  absence or change of periapical radiolucency is measured by standardized radiographs (paralleling technique every 3 months and cbct after 1 year)

SECONDARY OUTCOMES:
measuring different root parameters | 1 year
  using standardized radiographic assessment ( CBCT after 1 year and paralleling technique every 3 months for 1 year ) to assess
  1. Change in root length in millimeters
  2. Change in root thickness in millimeters
  3. Change in apical diameter in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Mai Abdel Raouf, Teaching assistant, Principal Investigator — Ainshams University
Locations (1):
- Faculty of Dentistry Ainshams University, Cairo, Egypt

REFERENCES:
- [Background] Dhillon H, Kaushik M, Sharma R. Regenerative endodontics--Creating new horizons. J Biomed Mater Res B Appl Biomater. 2016 May;104(4):676-85. doi: 10.1002/jbm.b.33587. Epub 2015 Dec 24. PMID 26699211